CLINICAL TRIAL: NCT06744543
Title: Randomized Controlled Trial to Assess EHR Prediction Model to Identify Pediatric Patients With Undiagnosed Genetic Disease"
Brief Title: Clinical Decision Support to Identify Pediatric Patients With Undiagnosed Genetic Disease
Acronym: SIGHT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Douglas Ruderfer, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 241678
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Genetic Disease; Pediatrics; Predictive Model; Clinical Decision Support
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Intervention Model Description: 1:1 allocation by predicted probability to either the intervention group, receiving a SIGHT-prompted provider message, or the control group, receiving standard care without the SIGHT-prompted message. The randomization process will be integrated into the routine clinical workflow, with SIGHT scores generated before regularly scheduled patient visits in pediatric primary care at VUMC.
Masking Description: There will be no blinding of participants or physicians as patients and providers will follow standard of care. Providers may dismiss the SIGHT - prompted provider message and not act on its recommendations at any time. No other intervention is planned. Patients would be unaware of the providers' decisions in that case unless the provider chooses independently to discuss the SIGHT score with them. A sample size re-estimation will be conducted after 250 patients have been randomized to account for uncertainty in the initial test-referral rate used in the sample size calculation. An independent analyst, who will be blinded to the randomization assignment, will calculate the observed test-referral rate across all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): SIGHT predictions will be generated prior to a scheduled encounter in one of the participating study clinics. Patients with a SIGHT probability above a predefined risk level (0.30 predicted risk based on validation and prior chart review by a genetic counselor, Morley et al, 2021 below) will prompt randomization to the standard care or SIGHT-guided intervention arm.
  For patients randomized to the SIGHT-guided intervention arm, the clinician responsible for care in that encounter (determined in the usual course of care) will receive a message for that patient and details as to the contributing clinical features that led to the high probability.
  The message will include a recommendation, but providers will have full discretion to offer genetic testing or refer to genetics providers. The management of screening will follow standard of care at VUMC.
  Interventions: Device: SIGHT Prompted Provider Message
- Comparator (No Intervention): All remaining patients will be the comparator arm which will be standard of care as to avoid ethical situations of withholding potentially important care.

INTERVENTIONS:
Device: SIGHT Prompted Provider Message — Among patients surpassing a 0.30 probability threshold that have a scheduled visit to pediatric primary care at VUMC, 500 will be randomized to the intervention and a SIGHT-prompted provider message will be generated.
  Arms: Intervention

SUMMARY:
This study will evaluate the effectiveness of SIGHT as a clinical support system to prompt provider/patient discussion and shared decision making regarding the need for genetic testing in the form of a chromosomal microarray. Identifying patients at high predicted probability of needing a test in clinical settings will be examined to determine if it decreases the duration of time to testing and increases diagnostic yield. SIGHT requires only data already collected in routine clinical encounters and is calculated prior to a clinical visit at VUMC.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 1 year old, < 20 years of age with a scheduled visit to the VUMC pediatric primary care.

Exclusion Criteria:

* Patients who have been programmatically excluded due to having already received a chromosomal microarray at VUMC and patients > 20 years of age or < 1 year of age.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Diagnoses in the intervention arm compared to the control arm | 2 years
  Number of patients diagnosed via a Chromosomal Microarray.

SECONDARY OUTCOMES:
Time to test | 2 years
  Duration of time to genetic testing. Time to event, measured from the initial patient visit to the time genetic testing is conducted.
Abnormal CMA | 2 years
  Number of patients flagged by SIGHT who's CMA result returned abnormal but in the absence of diagnostic findings.
Rate of genetic testing | 2 years
  Rates of genetic testing ordered by providers after a pediatric visit.
Diagnosis via any test (molecular confirmation) | 2 years
  Number of patients flagged by SIGHT who receive a diagnosis via any molecular test.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Ruderfer, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Patients in this study will receive standard of care at Vanderbilt University Medical Center (VUMC) and will not be consented for research participation. As a result, no individual participant data (IPD) will be made available for sharing with other researchers.

REFERENCES:
- [Background] Morley TJ, Han L, Castro VM, Morra J, Perlis RH, Cox NJ, Bastarache L, Ruderfer DM. Phenotypic signatures in clinical data enable systematic identification of patients for genetic testing. Nat Med. 2021 Jun;27(6):1097-1104. doi: 10.1038/s41591-021-01356-z. Epub 2021 Jun 3. PMID 34083811

DOCUMENTS (1):
  • Study Protocol (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT06744543/Prot_001.pdf